CLINICAL TRIAL: NCT05599620
Title: Reducing Alcohol Use and Sexual Dysfunction in Survivors of Sexual Trauma
Acronym: AWARE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lifespan (Other)
Responsible Party: Principal Investigator, Lindsay Orchowski Ph.D., Professor (Research), Lifespan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R34AA028402 (NIH)
Record Dates: First submitted 2022-10-25; First posted 2022-10-31 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Use, Unspecified; Sexual Dysfunction; Sexual Assault
MeSH Terms: conditions — Alcohol Drinking; Sexual Dysfunction, Physiological

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AWARE Program (Experimental): The AWARE program addresses alcohol use, sexual distress and sexual revictimization risk.
  Interventions: Behavioral: AWARE
- Control Group (No Intervention): The comparison is a wait list control group.

INTERVENTIONS:
Behavioral: AWARE — AWARE addresses alcohol use, sexual distress, and sexual assault risk among college women with a history of sexual victimization.
  Arms: AWARE Program

SUMMARY:
The goal of this clinical trial is to develop and evaluate the preliminary efficacy of an intervention to address alcohol use, sexual distress, and sexual assault risk among college women with a history of sexual victimization. The main questions it aims to answer are: 1) what is the feasibility of the recruitment method, research design, interventionist training methods, and delivery of the intervention; 2) does the intervention, relatively to control, the 2- and 4-month follow-up produces reductions in the quantity/frequency of alcohol use and heavy drinking, sexual distress, and sex-related drinking motives, and sexual revictimization. Participants will engage in both individual and group based intervention for alcohol use, sexual distress, and sexual assault risk. Follow-up assessments are completed at 2- and 4-months following program completion. The intervention is compared to a wait list control group who will have the opportunity to complete the program after completing the 4-month follow up.

ELIGIBILITY:
Inclusion Criteria:

1. be between the ages of 18 and 24;
2. speak and comprehend English;
3. report a history of attempted or completed penetrative or non-penetrative acts of sexual victimization (i.e., oral, vaginal, anal) since age 14 via incapacitation, coercion, or force;
4. report exceeding the national recommended limits for daily drinking (4 or more for women) on one or more occasions in the past 6 months;
5. report past year sexual activity;
6. exceed the clinical cut point on the Female Sexual Functioning Index (score of 28.1 or lower) or exceed the cut point for the 13-item Female Sexual Distress Scale-Revised (score of 11 or higher)

Exclusion Criteria:

1. suicide risk on items from the Beck Depression Inventory;
2. screen positive on the Alcohol Use Withdrawal Checklist.

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The intervention enrolls cis-gender college women.
Enrollment: 90 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Alcohol Use | Change from baseline alcohol use at 4 months.
  The number of past month drinking days (Minmum = 0, Maximum = 30), average drinks per drinking day (Minmum = 0, Maximum = unspecificed), number of heavy drinking days (Minimum = 0, Maximum = 30), assessed via the Time Line Follow Back, with greater scores meaning worse outcomes.
Sexual Distress | Change from overall levels of sexual dysfunction at 4 months.
  Assessed via the Female Sexual Dysfunction Index, Minimum = 2, Maximum = 36 with higher scores meaning worse outcomes, and the Female Sexual Distress Scale, Minimum = 0, Maximum = 52 with lower scores meaning worse outcomes.
Sexual Victimization | Reductions in severity and frequency of victimization in comparison to control at 4 months.
  Assessed via the Sexual Experiences Survey. Scored based on frequency and severity, Minumum = 0, Maximum = 63, higher scores means worse outcomes.

SECONDARY OUTCOMES:
Sex-Related Drinking Expectancies | Change in sexual related drinking expectancies at 4 months.
  Assessed via the Sex Related Alcohol Expectancies, Minimum = 14, Maximum = 70

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared using the National Institute of Mental Health Data Archive (NDA).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The research team will submit data on or before the NDA submission due dates (April 1 and October 1 each year) in accordance with the applicable Data Sharing Terms and Conditions of award.